CLINICAL TRIAL: NCT05800847
Title: Gabapentin Following Arthroscopic Rotator Cuff Repair: Evaluation of Postoperative Opioid Use and Sleep Quality
Brief Title: Effect of Gabapentin on Sleep and Opioid Use Following Rotator Cuff Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hughston Clinic (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HIRB2022-05
Record Dates: First submitted 2023-03-21; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Repair; Gabapentin; Opioid Use
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Patients in this arm will be receiving 100 mg placebo q8h for 2 days followed by 300 mg placebo q8h for 12 days. Patients will also receive 30 pills of hydrocodone-acetaminophen 5-325 mg q4-6h as needed.
  Interventions: Drug: Placebo
- Gabapentin (Experimental): Patients in this arm will be receiving 100 mg gabapentin q8h for 2 days followed by 300 mg gabapentin q8h for 12 days. Patients will also receive 30 pills of hydrocodone-acetaminophen 5-325 mg q4-6h as needed.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin will be administered for 2 days at 100 mg q8h for titration to avoid side effects. The next 12 days, gabapentin will be taken at 300 mg q8h.
  Arms: Gabapentin
Drug: Placebo — Placebo will follow the same dosing pattern as gabapentin to allow for blinding. Placebo will be encapsulated with a gelatin capsule to mimic the look of gabapentin.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effects of gabapentin in patients undergoing rotator cuff repair surgery. The main question it aims to answer is whether gabapentin can improve postoperative pain and sleep quality. Participants in this study will be randomized to either take gabapentin after surgery or a placebo after surgery.

DETAILED DESCRIPTION:
Perioperative gabapentin use has been established in prior literature to decrease postoperative opioid use; however, all of these studies have evaluated gabapentin given by an anesthesia team in the immediate pre- or intraoperative period. No known literature exists regarding scheduled post-operative oral gabapentin use in regards to pain control and opioid use. Sleep quality still tends to be a frequent concern associated with rotator cuff injury and shoulder surgery in general. The added known benefit of somnolence or drowsiness, in addition to aid in sleep, with use of gabapentin may also contribute to improved sleep quality following rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed traumatic or degenerative rotator cuff tear undergoing primary arthroscopic repair
* between the ages of 18 and 65 years old

Exclusion Criteria:

* chronic pre-operative narcotic pain medication use
* undergoing superior capsular reconstruction / balloon interposition etc
* < 18 y/o or > 65 y/o
* bilateral rotator cuff tear
* currently taking prescribed sleep-aid medications
* history of fibromyalgia or chronic pain syndrome
* pain management patient
* narcolepsy diagnosis
* diagnosis of cervical radiculopathy
* reported non-shoulder pain interfering with sleep

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Usage of Opioids for Pain Control | Up to 12 weeks postoperatively
  Determined based on morphine milligram equivalents
Change in Sleep Quality | Up to 12 weeks postoperatively
  Determined with Patient-Reported Outcomes Measurement Information System Sleep Disturbance Scale (min: 8, max: 40, higher score represents worse sleep)

SECONDARY OUTCOMES:
Change in Pain | Up to 12 weeks postoperatively
  Determined with Visual Analog Scale (min: 0, max: 10, higher score represents more pain)
Change in Functional Outcome (Based on Prior Baseline) | Up to 12 weeks postoperatively
  Determined with Single Assessment Numerical Evaluation (min: 0, max: 100, higher score represents better outcome)
Change in Functional Outcome (Based on Survey) | Up to 12 weeks postoperatively
  Determined with American Shoulder and Elbow Surgeons Scores (min: 0, max: 100, higher score represents better outcome)

IPD SHARING:
Plan to Share IPD: No